CLINICAL TRIAL: NCT00589485
Title: Total Knee Replacement Using Simplex® or Cobalt™ Bone Cement
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor did not fund the study
Sponsor: Zimmer Biomet (Industry)
Collaborators: New Lexington Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 102-U-012
Record Dates: First submitted 2007-12-21; First posted 2008-01-09 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Traumatic Arthritis; Knee Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
  Interventions: Device: Simplex® Bone Cement
- 2
  Interventions: Device: Cobalt™ Bone Cement

INTERVENTIONS:
Device: Simplex® Bone Cement — This arm will utilize Simplex® Bone Cement in total knee replacement.
  Groups: 1
Device: Cobalt™ Bone Cement — This arm utilizes Cobalt™ Bone Cement in total knee replacement.
  Groups: 2

SUMMARY:
The purpose of this study is to collect radiographic and clinical outcomes of total knee replacement using Simplex® or Cobalt™ Bone Cement.

DETAILED DESCRIPTION:
The purpose of this study is to collect radiographic and clinical outcomes of total knee replacement using Simplex® or Cobalt™ Bone Cement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with painful and disabled knee joint resulting from osteoarthritis, rheumatoid arthritis, traumatic arthritis where one or more compartments are involved
* Patients requiring correction of varus, valgus, or posttraumatic deformity
* Patients requiring correction or revision of unsuccessful osteotomy, arthrodesis, or failure of previous joint replacement procedure

Exclusion Criteria:

* Infection, sepsis, and osteomyelitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients who require total knee replacement.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-11; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Radiographic analysis and Knee Society Score | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Biomet Orthopedics, LLC, Warsaw, Indiana, United States